CLINICAL TRIAL: NCT05935969
Title: Endoscopic Transpapillary Gallbladder Drainage for Prevention of Biliary Complication in Surgically Unfit Patients With Both Choledocholithiasis and Cholecystolithiasis
Brief Title: ETGBD in Surgically Unfit Patients With Both Choledocholithiasis and Cholecystolithiasis
Acronym: ETGBD
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Hyun Paik, Associate Professor, Seoul National University Hospital
Other Study IDs: 2305-030-1429
Record Dates: First submitted 2023-06-27; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Efficacy
Keywords: Endoscopic transpapillary gallbladder drainage; High risk surgery; Gallstone; Common bile duct stone
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ERCP(Endoscopic retrograde choangiopancreatography), ETGBD(endoscopic transpapillary gallbladder drainage) — For transpapillary gallbladder drainage, biliary cannulation was performed with a duodenoscope (JF-260V or TJF-260V; Olympus Optical). After successful deep cannulation of the CBD, we checked the cholangiogram, performed endoscopic sphincterotomy, and removed the CBD stone using a memory basket and/or retrieval balloon. Cholangiography was then performed again to locate the cystic duct orifice, and a guide wire (Jagwire; Boston Scientific, Marlborough, Massachusetts, USA or Visiglide; Olympus, Tokyo, Japan) was inserted into the gallbladder with different types of catheters (standard catheter, pull-sphincterotome, or rotating sphincterotome) under fluoroscopic guidance. After placement of the guide wire into the gallbladder, contrast dye was injected to confirm good entry into the gallbladder. Once the gallbladder was selected and the guidewire was coiled in the GB, a 7Fr 12-15cm double pigtail plastic stent (Zimmon; Wilson-Cook Medical, Winston-Salem, NC) was inserted into the GB.

SUMMARY:
Cholecystectomy is recommended for patients with both gallbladder (GB) and common bile duct (CBD) stones to prevent recurrent biliary complications, unless there are specific reasons for surgery is considered inappropriate. The aim of this study was to evaluate the role of transpapillary gallbladder stent placement in surgically unfit patients with both CBD stone and gallstone.

DETAILED DESCRIPTION:
Gallstones affect 10-15% of the adult population, and 10-25% of them may develop biliary pain or complications. Patients with symptomatic gallstones often have a concomitant CBD stone in 10-20% of them. Most gallstones do not require invasive treatment due to their benign natural history, but CBD stones should be removed due to the risk of developing gallstone-related complications such as obstructive cholangitis and acute gallstone pancreatitis. CBD stones result mainly from the migration of gallstones into the bile duct, so the gold standard treatment for gallstones with CBD stones is endoscopic removal of the CBD stone followed by cholecystectomy to prevent recurrent biliary complications, such as calculous cholangitis or acute cholecystitis.

However, patients who were ineligible for surgery due to high-risk conditions, including the elderly, critically ill status, and severe underlying morbidities, may not get the chance to undergo cholecystectomy. Initial nonoperative management with delayed cholecystectomy has been considered as an alternative treatment, but laparoscopic cholecystectomy reduces the rate of major complications compared with percutaneous gallbladder drainage, even in high-risk patients, and outcomes after early laparoscopic cholecystectomy in octogenarians are comparable to younger patients. Despite this evidence, there are still debates among experts for optimal treatment methods for high-risk patients for surgery with symptomatic CBD stone with gallstone, and gallbladder drainage therapy first to perform for stabilization with surgery rather than urgent cholecystectomy in real practice. Therefore, there is still an unmet need for how to prevent recurrence of CBD stones in patients with concomitant gallstones after endoscopic removal of CBD stones.

Nonsurgical cholecystic drainage methods, including percutaneous transhepatic gallbladder drainage (PTGBD), endoscopic ultrasound-guided gallbladder drainage (EUS-GBD), and endoscopic transpapillary gallbladder drainage (ETGBD), have been introduced and actively used as a bridge or alternative therapy in patients at high risk for surgery. Several studies have reported the results of its feasibility and efficacy, mainly focusing on the management of patients with acute cholecystitis. However, the evidence for appropriate management considering non-surgical treatments for patients with both CBD stones and gallstones is still limited. This study evaluated the feasibility and efficacy of ETGBD for patients with both CBD stone and gallstones to prevent recurrent biliary complications in patients at high risk for surgery.

ELIGIBILITY:
Inclusion Criteria:

(i) age ≥20 years (ii) presence of choledocolithiasis and cholecystolithiasis on imaging studies (iii) surgically unfit for cholecystectomy.

Exclusion Criteria:

(i) presence of malignant biliary obstruction (ii) follow-up of less than 1 month (iii) previous EST status (iv) pregnancy

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: From January 2010 to March 2022, 302 patients with both choledocholithiasis and cholecystolithiasis who were at high surgical risk, were reviewed retrospectively. All 302 patients were initially treated with endoscopic CBD stone removal.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Recurrence of biliary complications | through study completion, an average of 2 year
  The primary outcome measures were biliary complications, including acute cholecystitis, acute cholangitis, recurrence of choledocolithiasis, and biliary colic. The diagnosis of acute cholangitis, acute cholecystitis were based on Tokyo guideline 18.

CONTACTS AND LOCATIONS:
Overall Officials: Myeong Hwan Lee, M.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Due to the sensitive nature of the subject of this work and also the clinical data used, our healthboard stipulates that raw data should remain confidential and not be shared.

REFERENCES:
- See also: pubmed — http://pubmed.ncbi.nlm.nih.gov/advanced/